CLINICAL TRIAL: NCT02858063
Title: Psychometric Validation of a Subjective Quality-of-life Scale in Young Women With a Non Metastatic Breast Cancer and Her Partner (KALICOU 2 Protocol)
Brief Title: Psychometric Validation (Quality-of-life Scale) in Young Women With a Non Metastatic Breast Cancer and Her Partner
Acronym: KALICOU2
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Université Lille 3 (Unknown)
Responsible Party: Sponsor
Other Study IDs: KALICOU2-0909
Record Dates: First submitted 2016-08-03; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Quality Of Life; Women; Partner
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pending chemotherapy +/- trastuzumab: In the 1st group (chemotherapy), 25 couples will answer to kalicou questionnaire (KALI), 25 couples to KALI plus QLQC-30 and QLQBR-23 questionnaires for patients and SF-36 questionnaire for their partners. 25 couples will answer to KALI plus STAI plus CES-D questionnaires and 25 couples will ansmwer twice to KALI questionnaire, with a delay of 15 days between each other
- pending trastazumab +/- hormone therapy: In the 2nd group (trastazumab), 25 couples will answer to kalicou questionnaire (KALI), 25 couples to KALI plus QLQC-30 and QLQBR-23 questionnaires for patients and SF-36 questionnaire for their partners. 25 couples will answer to KALI plus STAI plus CES-D questionnaires and 25 couples will ansmwer twice to KALI questionnaire, with a delay of 15 days between each other
- pending hormone therapy alone: In the third group (hormone therapy), 25 couples will answer to kalicou questionnaire (KALI), 25 couples to KALI plus QLQC-30 and QLQBR-23 questionnaires for patients and SF-36 questionnaire for their partners. 25 couples will answer to KALI plus STAI plus CES-D questionnaires and 25 couples will ansmwer twice to KALI questionnaire, with a delay of 15 days between each other
- pending afercare period: In the last group (aftercare), 25 couples will answer to kalicou questionnaire (KALI), 25 couples to KALI plus QLQC-30 and QLQBR-23 questionnaires for patients and SF-36 questionnaire for their partners. 25 couples will answer to KALI plus STAI plus CES-D questionnaires and 25 couples will ansmwer twice to KALI questionnaire, with a delay of 15 days between each other

SUMMARY:
* Selection of patient and preparation of questionnaires
* Presentation of the study by the doctor
* Verbal consent of participants (patient and Partner)
* Delivery of booklets
* Response to documents (questionnaires and written consent) at home, send by mail

DETAILED DESCRIPTION:
1. Before consultation :

   Selection of patients according to inclusion criteria by persons in charge and preparation of inclusion file
2. During the consultation :

   * Presentation of the study by the investigator
   * The investigator signs the information note and give two file to the patient (1 for her and 1 for her Partner : both contains 1 information note signed by the investigator, 1 questionnaire and 2 stamped envelopes
   * Finally, the investigator fill-in the medical form and send the original to the university (université de Lille 3)
3. At home :

   * Signature of the information note and the participation consent form
   * Patients and Partner responds to their questionnaire (including socio-demographique questionnaire)
   * They send the documents thanks to stamped envelopes:

     1. They send information note to the medical center
     2. They send the questionnaires to the university

ELIGIBILITY:
Inclusion Criteria:

* >18 years old (patient and partner)
* <45 years old (patient)
* Patient with a non metastatic breast cancer
* Patient treated or previously treated by chemotherapy
* Patient and her Partner live together for at least 6 months when they complete the questionnaires.

Exclusion Criteria:

* Patient or patner with psychiatric trouble
* Native language other than french

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young women (<45 years old)treated or previously treated by chemotherapy for a non metastatic breast cancer, in Relationship for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 1045 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
psychometric validation of a questionnaire in Young patients and their partners | 1 year

SECONDARY OUTCOMES:
compare convergent and or divergent dimensions with patients and theirs partners | 1 year
compare responses of participants according to traitement/ surveillance period | 1 year

IPD SHARING:
Plan to Share IPD: No